CLINICAL TRIAL: NCT03910751
Title: Project to Look for Early Discharge in Patients Undergoing TAVI With ACURATE - An International Multi-center Early Discharge TAVI Program
Brief Title: POLESTAR Trial - An International Multi-center Early Discharge TAVI Program
Acronym: POLESTAR
Status: Completed | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Principal Investigator, Nicolas van Mieghem, Principal Investigator, Erasmus Medical Center
Other Study IDs: POLESTAR_EMC2019
Record Dates: First submitted 2019-03-26; First posted 2019-04-10 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-06

CONDITIONS: Aortic Valve Stenosis
Keywords: TAVI; TAVR; Early discharge; ACURATE Neo
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Transcatheter Aortic Valve Implantation with ACURATE Neo Aortic Bioprosthesis — Transfemoral TAVI using the Boston Scientific ACURATE Neo Aortic Bioprosthesis

SUMMARY:
An international multi-center prospective observational study to address safety and feasibility of an early discharge protocol in patients with symptomatic severe aortic stenosis who are eligible for transfemoral TAVI with the Boston Scientific ACURATE Neo Aortic Bioprosthesis transcatheter heart valve.

DETAILED DESCRIPTION:
In this International multi-center prospective observational study, 250 patients with severe symptomatic aortic stenosis (AS) and eligibility for transfemoral TAVI with ACURATE Neo Bioprosthesis, will be pre-procedurally selected for participation in an early discharge protocol in which patients are discharged within 48 hours after uncomplicated TAVI.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for ACURATE Neo valve implantation
* Patient agrees to follow-up duration
* Patient is able to understand and sign written informed consent

Exclusion Criteria:

* BMI > 35
* Pregnancy

Cardiac

* Moderate to severely impaired left ventricular ejection fraction (LVEF <35%)
* Mitral regurgitation > moderate
* Pulmonary hypertension (sPAP > 60mmHg)
* No complex coronary artery disease
* Untreated high degree AV-block or RBBB

Pulmonary

* COPD Gold > 2

Kidney function

* GFR < 35ml/min

Frailty

* Inappropriate social support and/or (familial) care
* Patient is walking aid dependent

TAVI strategy

* Presence of severe peripheral artery disease
* Transfemoral approach not possible

Follow up

* Inability to adhere to follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 250 patients with severe AS and selected for TF-TAVI with the ACURATE Neo valve and eligible for early discharge within 48 hours post TAVI
Sampling Method: Non-Probability Sample
Enrollment: 252 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2022-12-05 (Actual); Study Completion 2024-01-24 (Actual)

PRIMARY OUTCOMES:
Primary safety endpoint | 30 days
  Composite of all-cause mortality, any stoke, VARC type 2-4 bleeding, acute kidney injury stage 3-4, major vascular, major access related, major cardiac structural complication, moderate or severe aortic regurgitation, new permanent pacemaker implantation and valve-related dysfunction requiring repeat procedure at 30 days
Primary efficacy endpoint at 30 days | 30 days
  Composite of all-cause mortality, all stroke, re-hospitalization for procedure- or valve-related causes, KCCQ Overall Summary Score <45 or decline from baseline >10 points at 30 days
Primary efficacy endpoint at 1 year | 1 year
  Composite of all-cause mortality, all stroke, re-hospitalization for procedure- or valve-related causes, KCCQ Overall Summary Score <45 or decline from baseline >10 points at 1 year

SECONDARY OUTCOMES:
All-cause mortality | 30 days and 1 year
  As defined by the most recent VARC document
Stroke | 30 days and 1 year
  As defined by the most recent VARC document
Life threatening bleeding | 30 days and 1 year
  As defined by the most recent VARC document
Acute kidney injury | 30 days and 1 year
  As defined by the most recent VARC document
Coronary artery obstruction requiring intervention | 30 days and 1 year
  As defined by the most recent VARC document
Major vascular complication | 30 days and 1 year
  As defined by the most recent VARC document
Valve related dysfunction requiring repeat procedure | 30 days and 1 year
  As defined by the most recent VARC document
All-cause rehospitalization | 30 days and 1 year
  As defined by the most recent VARC document
Rehospitalization for valve-related symptoms or worsening congestive heart failure | 30 days and 1 year
  As defined by the most recent VARC document
New permanent pacemaker implantation | 30 days and 1 year
  As defined by the most recent VARC document
Myocardial infarction | 30 days and 1 year
  As defined by the most recent VARC document
NYHA heart failure class III or IV | 30 days and 1 year
  As defined by the most recent VARC document
Patient reported Quality of Life | 30 days and 1 year
  As measured by the EQ5D-5L quality of life questionnaire
Patient reported Quality of Life | 30 days and 1 year
  As measured by the KCCQ quality of life questionnaire
Categorical cost analysis | 30 days
  Derived from length of stay on Intensive care unit and general ward

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Van Mieghem, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (15):
- Belgium (4):
  - ASZ Aalst, Aalst
  - AZ Sint-Jan Brugge, Bruges
  - UZ Brussel, Brussels
  - AZ Maria Middelares, Ghent
- Canada (3):
  - Royal Columbian Hospital, New Westminster
  - Sunnybrook Health Sciences Centre, Toronto
  - Vancouver General Hospital, Vancouver
- Netherlands (5):
  - University Medical Center Groningen, Groningen
  - Leiden University Medical Center, Leiden
  - St. Antonius Hospital, Nieuwegein
  - Erasmus University Medical Center, Rotterdam
  - Utrecht University Medical Center, Utrecht
- United Kingdom (3):
  - University Hospital Sussex NHS Foundation Trust, Brighton
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - University Hospitals of Leicester NHS Trust, Leicester

IPD SHARING:
Plan to Share IPD: Undecided